CLINICAL TRIAL: NCT03985904
Title: Museum-based Group Art Therapy in the Process of Mental Health Recovery and Spanish Cultural Adaptation and Validation of the Questionnaire About the Process of Recovery (QPR-15)
Brief Title: Museum-based Group Art Therapy in Mental Health Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: University of Alcala (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0385-N-19
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-02

CONDITIONS: Psychosis
Keywords: mental health recovery; art therapy; museum
MeSH Terms: conditions — Psychotic Disorders | interventions — Art Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Art Therapy (Experimental): Participants will attend art therapy group sessions for three months in a designated museum.
  Interventions: Other: ART THERAPY

INTERVENTIONS:
Other: ART THERAPY — ART THERAPY: Nursing Interventions Classification = 4330 Weekly 2 hour group carried out by a mental health nurse, a social monitor and a museum educator.

SUMMARY:
This clinical trial aims to evaluate the effects of an art therapy intervention carried out in museums to facilitate the process of recovery in mental health. In total 100 users of mental health services will be recruited for this study. Participants in the trial will be assessed at baseline and at 3 months.

DETAILED DESCRIPTION:
Art therapy

QUALITY ASSURANCE PLAN. The researchers will review and report the process during the trial covering participant enrolment, consent and eligibility to protect participants, including reporting of harm and completeness, accuracy and timeliness of data collection.

STANDARD OPERATING PROCEDURES. Participants will be recruited over a period of three months by mental health professionals (mental health nurses, psychologists, psychiatrists and occupational therapists). Participants will not receive financial reimbursement for taking part in this trial. Participants will be identified from outpatient services who meet all the study eligibility criteria (listed in section Eligibility). ICD-10 (International Classification of Diseases) and GAF (Global Assessment of Functioning) will be used to screen participants at recruitment.

DATA DICTIONARY. All variables collected in this study will be listed and described in a case report form, with associated guidelines, to ensure consistency in all gathered data. The following data will be collected in this trial:

Sociodemographical data Clinical history Global Assessment of Functioning Scale (GAF) Questionnaire about the Process of Recovery (QPR-15) Visual Analogue Recovery Scale Duke-UNC Functional Social Support Questionnaire

SAMPLE SIZE ASSESSMENT. The estimated sample size is n = 102, for a t test with two independent samples, with one tail, an effect size of 0.5, an α of 95% and a power of 80%.

For the validation of the QPR-15, taking into account the subject-item ratio of at least 5: 1 (15 items), and considering the minimum number of recommended subjects to perform an Exploratory Factor Analysis, The minimum number of participants must be 100.

Thus, estimating losses of 20%, the total number of participants estimated for the study is n = 127.

STATISTICS ANALYSIS PLAN. The change of means in the main outcome variable will be analyzed with the Student's t-test and if the criteria for its application with the nonparametric Mann-Whitney U test are not met. For the categorical secondary variables, the Chi square test will be used.For all comparisons, a confidence level of 95% will be used. The program R version 3.5.1 will be used. for all statistical analyzes.

PLAN FOR MISSING DATA. Each researcher is responsible for ensuring that any missing data will be reported as missing in the study database. Procedures can sometimes be considered when using statistical methods that fail in the presence of any missing values, or when in the case of multiple-predictor statistical models all the data for an individual would be omitted because of a missing value in one of the predictors. For analyzes involving multiple regression analysis, a multiple imputation approach will be considered and used if statistically sound, depending on the proportion and pattern of missing values.

METHODS TO ENSURE VALIDITY AND QUALITY OF DATA. Accurate and reliable data collection will be assured by verification and cross-check of the case report form (CRF) against the researcher´s records (source document verification). Source document verification will be conducted for 5% of data in subjects. Discrepancies and queries will be generated accordingly in the CRF for online resolution by the researcher at the site. In addition, the CRF data will be reviewed on an ongoing basis for medical and scientific plausibility.

ELIGIBILITY:
Inclusion Criteria:

* Participants are 18 years or older.
* Participants have a diagnosis of ICD-10 F20-29 or F31.7 with a psychotic history.
* Participants agree to be part of the study by giving signed written consent.

Exclusion Criteria:

* Score in GAF <50 points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline personal recovery in adults in mental health follow-up at 3 months. | At baseline then at 3 months.
  Questionnaire about the Process of Recovery (QPR-15) is an instrument of 15 items to measure the recovery of people using mental health services. Each item is scored using a Likert-type scale of 0 (strongly disagree) to 4 (strongly agree) with a total score of 0 to 60.

SECONDARY OUTCOMES:
Change from baseline social support in adults in mental health follow-up at 3 months. | At baseline then at 3 months.
  Duke-UNC Functional Social Support Questionnaire is a self-administered questionnaire of 11 items to measure perceived social support. Each item is scored using a Likert-type scale of 1 (much less than I would like) to 5 (as much as I would like) with a score ranging between 11 and 55 points. In the Spanish validation, a cut point was chosen in the 15th percentile, which corresponds to a score lower than 32 indicating a low perceived social support and a score equal to or greater than 32 indicating a normal support.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Goodman Casanova, Principal Investigator — IBIMA - FIMABIS
Locations (1):
- Jessica Marian Goodman Casanova, Málaga, MA, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Law H, Neil ST, Dunn G, Morrison AP. Psychometric properties of the questionnaire about the process of recovery (QPR). Schizophr Res. 2014 Jul;156(2-3):184-9. doi: 10.1016/j.schres.2014.04.011. Epub 2014 May 9. PMID 24816049
- [Background] Moorhead S, Johnson M, Maas ML, Swanson E. Clasificación de Resultados de Enfermería (NOC). Elsevier España, S.L. 2013.
- [Background] Bellon Saameno JA, Delgado Sanchez A, Luna del Castillo JD, Lardelli Claret P. [Validity and reliability of the Duke-UNC-11 questionnaire of functional social support]. Aten Primaria. 1996 Sep 15;18(4):153-6, 158-63. Spanish. PMID 8962994
- [Background] Servicio Andaluz de Salud. Escala de evaluación global de funcionamiento o Escala de evaluación de la actividad global (EEAG) Global Assessment of Functioning Scale (GAF). 2010; Disponible en: http://www.juntadeandalucia.es/servicioandaluzdesalud/contenidos/publicaciones/Datos/433/pdf/14-GAF.pdf
- [Background] Chisholm D, Knapp MR, Knudsen HC, Amaddeo F, Gaite L, van Wijngaarden B. Client Socio-Demographic and Service Receipt Inventory--European Version: development of an instrument for international research. EPSILON Study 5. European Psychiatric Services: Inputs Linked to Outcome Domains and Needs. Br J Psychiatry Suppl. 2000;(39):s28-33. doi: 10.1192/bjp.177.39.s28. PMID 10945075
- [Background] Ruddy R, Milnes D. Art therapy for schizophrenia or schizophrenia-like illnesses. Cochrane Database Syst Rev. 2005 Oct 19;2005(4):CD003728. doi: 10.1002/14651858.CD003728.pub2. PMID 16235338
- [Background] Attard A, Larkin M. Art therapy for people with psychosis: a narrative review of the literature. Lancet Psychiatry. 2016 Nov;3(11):1067-1078. doi: 10.1016/S2215-0366(16)30146-8. Epub 2016 Aug 12. PMID 27528095